CLINICAL TRIAL: NCT05786586
Title: Repeated Exposure to 650nm Low-level Red-light for Myopia Control and Prevention in Children: a Randomized Controlled Trial
Brief Title: 650nm Low-level Red-light for Myopia Control and Prevention in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Children's Hospital (Other); Children's Hospital of The Capital Institute of Pediatrics (Other)
Responsible Party: Principal Investigator, Ying Jie, MD, Prof, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TongrenJY2022
Record Dates: First submitted 2023-01-29; First posted 2023-03-27 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 650 nm low-level red-light, plus single vision spectacle lenses (Experimental): Children in the treatment group are expected to receive 6 minutes irradiation of 650 nm low-level red-light daily, divided into two times a day, each lasting for 3 minutes. Single vision spectacle lenses are allowed for myopic children.
  Interventions: Device: 650 nm low-level red-light
- Control (No Intervention): Single vision spectacle lenses are allowed for myopic children. No intervention was given.

INTERVENTIONS:
Device: 650 nm low-level red-light — 650 nm low-level red-light is a kind of laser, concentrated into a beam, to repeatedly irradiate the retina
  Arms: 650 nm low-level red-light, plus single vision spectacle lenses

SUMMARY:
A multicenter randomized controlled trial, evaluating the efficacy and safety of 650nm low-level red-light irradiation for myopia control and prevention in children. Participants included children(aged 6 to 12 years, spherical equivalent error of 0.5D or below) who are already myopic at recruitment, and those who are of Emmetropia or low hyperopia.

DETAILED DESCRIPTION:
This multicenter randomized controlled trial will be conducted in three hospitals: Beijing Tongren Hospital, and another two subcenters. The whole study will last for five years.The investigators will perform data analysis at 6 months follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up and the end of the study. The intervention measure used will be 650 nm low-level red-light. This kind of intervention will be integrated into a headworn device. This device could be used for treatment of myopia or amblyopia, and is safe for the eyes and has been verified by the Chinese market supervision and administration department.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years
* The cycloplegic spherical equivalent error (SER) is -6D to 1D (> -6D, ≤1D) in both eyes
* Astigmatism of 2.5 D or less (≤2.5D)
* Willing to participate in the study and sign the informed consent form

Exclusion Criteria:

* Using other myopia interventions or stopped using them for less than three months, including but not limited to atropine eye drops or orthokeratology lens
* With anisometropia (difference in sphere between two eyes was 1.5D or greater), strabismus, or amblyopia
* With refractive media opacification (keratopathy, lens opacity, etc.)
* Allergy to cycloplegia drugs

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 572 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in axial length | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an optical biometer to measure the axial length.
Change in spherical equivalent error | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Children's pupil were dilated using Mydrin-P eye drops, and then the refractive error was measured using an autorefractor. the two measurements (axial length and spherical equivalent error) will be aggregated to arrive at one reported value through the following way: axial enlongation will be defined as progress in myopia, decrease in spherical equivalent error will be defined as progress in myopia too.

SECONDARY OUTCOMES:
Change in Choroid thickness | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an enhanced-depth imaging technique (based on Optical coherence tomography )
Change in steep keratometry | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an optical biometer
Change in flat keratometry | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an optical biometer
Change in length thickness | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an optical biometer
Change in anterior chamber depth | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an optical biometer
Change in central corneal thickness | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Use an optical biometer

OTHER OUTCOMES:
Fundus injury related to 650 nm low-level red-light irridiation | Baseline, six-month follow-up, one-year follow-up, two-year follow-up, three-year follow-up, four-year follow-up, five-year follow-up
  Any potential fundus injury related to 650 nm low-level red-light irridiation would be checked through Fundus photography and coherence tomography examination

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jie, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No